CLINICAL TRIAL: NCT07273617
Title: Effects of Positive End-Expiratory Pressure (PEEP) and Prone Positioning in Healthy Volunteers on Venous Hemodynamics Including the Venous Excess Ultrasound (VExUS) Score
Acronym: VeNIVPro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: am25Loosen2; 2025-01745
Record Dates: First submitted 2025-11-14; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Venous Hemodynamics
Keywords: Positive End-Expiratory Pressure (PEEP); Venous Excess Ultrasound (VExUS) score; Venous congestion; Proning
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Intervention Model Description: Prospective explorative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Supine position 2. Prone Position (Experimental): First body position: randomized to supine position. Randomization of starting PEEP (0 or 15 mbar) in first body position and sequence of measurements.
  Second body position: Prone Position. Randomization of starting PEEP (0 or 15 mbar) in second body position and sequence of measurements.
  Interventions: Diagnostic Test: application of PEEP: starting PEEP = 15 mbar; Diagnostic Test: application of PEEP: starting PEEP = 0 mbar
- 1. Prone Position 2. Supine Position (Experimental): First body position: randomized to prone position. Randomization of starting PEEP (0 or 15 mbar) in first body position and sequence of measurements.
  Second body position: Supine Position. Randomization of starting PEEP (0 or 15 mbar) in second body position and sequence of measurements.
  Interventions: Diagnostic Test: application of PEEP: starting PEEP = 15 mbar; Diagnostic Test: application of PEEP: starting PEEP = 0 mbar

INTERVENTIONS:
Diagnostic Test: application of PEEP: starting PEEP = 15 mbar — The application of PEEP will be delivered by a intensive care respirator with dedicated NIV- mode (Hamilton C1, Hamilton Medical AG, Bonaduz Switzerland) via mask (VariFit, Sleepnet Corporation, New Hampshire, USA) available in four sizes (S, M, L, XL). Pressure support will be set at 5 mbar, and trigger will be adjusted according to participants' comfort. Fraction of inspired oxygen will be 0.21. If starting PEEP = 15 mbar:
  5 min stepwise increase of PEEP Measurements with decremental PEEP (15, 10, 5, 0 mbar)
Diagnostic Test: application of PEEP: starting PEEP = 0 mbar — The application of PEEP will be delivered by a intensive care respirator with dedicated NIV- mode (Hamilton C1, Hamilton Medical AG, Bonaduz Switzerland) via mask (VariFit, Sleepnet Corporation, New Hampshire, USA) available in four sizes (S, M, L, XL). Pressure support will be set at 5 mbar, and trigger will be adjusted according to participants' comfort. Fraction of inspired oxygen will be 0.21. If starting PEEP = 0 mbar: Measurement with increasing PEEP (0, 5, 10, 15 mbar)

SUMMARY:
The hemodynamic effects of proning and PEEP may vary depending on pre- existing cardiac function, lung mechanics, and volume status, and the available evidence remains conflicting. The impact on the VExUS score of these manoeuvres is unclear. This study aims to assess the effects of PEEP in supine and prone position on the VExUS score as well as echocardiographic parameters in a cohort of healthy volunteers.

DETAILED DESCRIPTION:
Venous congestion: characterized by elevated venous pressure and impaired flow through the organs towards the right heart, contributes to organ dysfunction and is associated with adverse outcomes in critically ill patients. Historically, hemodynamic assessment has focused on the arterial side of circulation, giving less attention to venous hemodynamics. However, there is growing evidence that venous congestion is a mediator of adverse outcomes and contributes to end-organ damage. With increasing venous congestion, subsequent venous distension in the splanchnic circulation occurs and the pressure waveform of the right atrium is retrogradely transmitted into the distal venous circulation. The more venous congestion is present, the more pulsatility is transmitted into the periphery. This represents the backbone of the venous excess ultrasound (VExUS) score assessment. The VExUS score assessment therefore represents a multi-organ Doppler approach evaluating venous congestion by measuring the inferior vena cava (IVC) diameter, flow pattern of hepatic veins, portal vein and intra-renal veins by ultrasound.

Heart lung interactions and implications on VExUS: the VExUS score as well as femoral and jugular vein flows are expected to be affected by positive pressure ventilation. The VExUS score correlates with the Mean systemic filling pressure (MSFP) as a surrogate for stressed volume, in other words the proportion of blood which contributes to creating pressure and blood flow. As right atrial pressure is influenced by Positive End-Expiratory Pressure (PEEP), one would expect elevated VExUS Scores with higher PEEP levels.

Influence of position on hemodynamics: conflicting effects on the circulatory system mediated by prone positioning have been described; no data about VExUS Score assessment in prone position is available.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participants ≥ 18 years in good overall health with no relevant organ dysfunction in their medical history and signed informed consent form.

Exclusion Criteria:

* Non-French or non-German speakers
* Unable to provide informed consent
* Body mass index > 40kg/m
* Self-reported pregnancy
* History of pneumothorax
* Previously participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in VExUS score at 0, 5,10 and 15 mbar during non-invasive ventilation (NIV) in the supine position. | up to 15 min
  The Venous excess ultrasound (VExUS) score is a grading system that uses ultrasound to non-invasively assess and quantify systemic venous congestion by evaluating the inferior vena cava, hepatic veins, portal veins, and renal veins. A patient receives a grade from 0 (no congestion) to 3 (severe congestion) based on findings like IVC diameter and Doppler waveforms from the veins.

SECONDARY OUTCOMES:
Change in VExUS score at 0, 5,10,15 mbar during non-invasive ventilation in the prone position compared to the supine position. | up to 15 min
  The Venous excess ultrasound (VExUS) score is a grading system that uses ultrasound to non-invasively assess and quantify systemic venous congestion by evaluating the inferior vena cava, hepatic veins, portal veins, and renal veins. A patient receives a grade from 0 (no congestion) to 3 (severe congestion) based on findings like IVC diameter and Doppler waveforms from the veins.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Loosen, Dr. med., Principal Investigator — University Hospital Basel, Intensive Care Unit
Locations (1):
- University Hospital Basel, Intensive Care Unit, Basel, Switzerland